CLINICAL TRIAL: NCT06868680
Title: Prospective, Balance Program Study With Comparison Group
Brief Title: A Digital Balance Program With Comparison Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hinge Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20240129
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Falls
Keywords: balance; falls prevention; older adults; exercise therapy; telerehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Program (Experimental): A digital program of exercise therapy, access to physical therapist and health coach, and educational articles on falls prevention.
  Interventions: Behavioral: Balance Program
- Comparison Group (Active Comparator): Shared educational content on falls prevention and the importance of balance.
  Interventions: Other: Educational Reading Content

INTERVENTIONS:
Behavioral: Balance Program — A comprehensive program of tailored exercise therapy, educational content spanning a variety of topics related to balance improvement and fall prevention, a personalized clinical approach to improving balance, and access to a board-certified health coach and physical therapist.
  Arms: Balance Program
Other: Educational Reading Content — Informational articles on reducing risk for falls.
  Arms: Comparison Group

SUMMARY:
This research study evaluates a digital musculoskeletal care program specifically focused on balance improvement and falls prevention. The primary goal is to determine if the program results in fewer falls compared to a comparison condition where people will get educational/information articles on falls prevention. Study participants are asked to participate in their assigned condition and complete surveys throughout the study.

DETAILED DESCRIPTION:
The digital Balance Program is accessible through a smartphone or tablet and includes tailored exercise therapy, educational content spanning a variety of topics related to balance improvement and fall prevention, a personalized clinical approach to improving balance, and access to a board-certified health coach and physical therapist. The comparison group consists of a series of emailed articles on falls prevention. In addition to participating in the assigned condition, participants are asked to answer surveys that ask questions related to your balance, mental health, demographic information, and lifestyle. The surveys are sent before, during and at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* had an email account and owned a smartphone
* had a moderate-high fall risk based on the Stopping Elderly Accidents, Deaths, and Injuries (STEADI) questionnaire (≥ 4 points)

Exclusion Criteria:

* undergone musculoskeletal surgery within three months prior to recruitment
* a history of opioid, alcohol, or drug abuse within the last year
* a diagnosis of cognitive, behavioral, neurologic, or psychiatric disorders
* any contraindication for light physical activity as directed by the prospective participant's doctor

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 687 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Annualized fall rate | 3 months
  Annualized fall rate was calculated at baseline as the total number of falls experienced within the past year, divided by 12. Annualized fall rate was calculated at month three as the total number of falls participants reported experiencing between baseline and month three, divided by 0.25 person-years

SECONDARY OUTCOMES:
Fall Severity | baseline to 3 months
  How severe was the worst fall you experienced: none, minor, moderate, major

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Castro Sweet, PhD, Study Director — Hinge Health, Inc
Locations (1):
- Hinge Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data are available from the study contact upon reasonable request